CLINICAL TRIAL: NCT00375609
Title: Evaluation of the Factor Xa Inhibitor, PRT054021, Against Enoxaparin in a Randomized Trial for the Prevention of Venous Thromboembolic Events After Unilateral Total Knee Replacement (EXPERT)
Brief Title: Factor Xa Inhibitor, PRT054021, Against Enoxaparin for the Prevention of Venous Thromboembolic Events (EXPERT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Portola Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Alexion Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRT05-003
Record Dates: First submitted 2006-09-11; First posted 2006-09-13 (Estimated); Results first posted 2017-12-15 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Thromboembolism
Keywords: Prevention of Venous Thromboembolism
MeSH Terms: conditions — Thromboembolism | interventions — betrixaban; Enoxaparin

ARMS (3):
- Betrixaban 15 mg (Experimental): Betrixaban 15 mg oral twice daily for 10 to 14 days
  Interventions: Drug: Betrixaban
- Betrixaban 40 mg (Experimental): Betrixaban 40 mg oral twice daily for 10 to 14 days
  Interventions: Drug: Betrixaban
- Enoxaparin (Experimental): Enoxaparin 30 mg administered subcutaneously every 12 hours for 10 to 14 days
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Betrixaban — Capsule
  Arms: Betrixaban 15 mg; Betrixaban 40 mg
Drug: Enoxaparin — Administered subcutaneously
  Other Names: Lovenox
  Arms: Enoxaparin

SUMMARY:
Randomized study of PRT054021 40 mg and 15 mg bid vs. enoxaparin 30 mg q12h for the prophylaxis of venous thromboembolic events after unilateral knee replacement surgery.

DETAILED DESCRIPTION:
Approximately 200 patients undergoing unilateral knee replacement will be entered into the study and randomized to receive either enoxaparin 30 mg sq bid, PRT054021 15 mg po bid, or PRT054021 40 mg po bid for 10 to 14 days, at which time patients will undergo venography.

ELIGIBILITY:
Inclusion Criteria:

* • The subject has undergone elective primary unilateral TKR (not unicompartmental).

Demographic

* The subject is between the ages of 18 and 75 years.
* If the subject is a woman, she is without reproductive potential (postmenopausal for >2 years or after hysterectomy).
* The subject weighs between 50 kg (110 lbs) and 120 kg (265 lbs). Laboratory and Procedures
* The subject is willing and able to undergo unilateral venography. Medications
* The subject is willing and able to self-inject enoxaparin or receive injections q12h by a caregiver.

Ethical • The subject is able to read and give written informed consent and has signed an informed consent form approved by the Investigator's IRB/IEC.

Exclusion Criteria:

* Disease Related

  * Major medical and/or surgical condition which may impair oral drug absorption or metabolism.
  * Immobilization for 3 or more days before surgery.
  * History (including family history) or symptoms of a congenital or acquired bleeding disorder or vascular malformation; or a history of intracranial, retroperitoneal, or intraocular bleeding within the last 6 months; or is felt to be at high risk for bleeding for other reasons.
  * Gastrointestinal bleeding within 90 days before surgery or endoscopically verified ulcer disease within 30 days before surgery.
  * Indwelling intrathecal or epidural catheter during the prophylaxis period (except for epidural catheter if removed after surgery); or unusual difficulty in administering spinal or epidural anesthesia (eg, 3 or more attempts, "traumatic taps").
  * Major surgery, ischemic stroke, or myocardial infarction within 3 months before Screening.
  * Uncontrolled hypertension defined as systolic blood pressure (SBP) > 180 mmHg or diastolic blood pressure (DBP) >105 mmHg.
  * Hypotension defined as SBP <95 mmHg.
  * Evidence at Screening of symptomatic congestive heart failure requiring treatment.
  * Chronic atrial fibrillation treated with oral anticoagulants, recurrent atrial arrhythmia(s) or a history of recurrent ventricular tachycardia.

Laboratory and Procedures

• Evidence at Screening of: platelet count <100,000/mm3 potassium <3.5 mEq/L hemoglobin concentration <10 g/dL or hematocrit <30% serum ALT or AST >2 times ULN serum creatinine >2.0 mg/dL (180 µm/L)

* Contraindication to venography, including to iodinated contrast medium
* QTc on Screening ECG >450 msec and/or a personal or family history of "Long QT Syndrome".

Medications

* Contraindication to anticoagulation for VTE prophylaxis, including a contraindication to receiving heparin or heparinoids.
* Administration of the following drugs within 7 days before TKR: thrombolytic agents, anticoagulants and/or anti-platelet agents (eg, heparins, warfarin, dipyridamole, sulfinpyrazone, ticlopidine, dextran, clopidogrel). Aspirin up to 325 mg once daily and NSAIDs are allowed but discouraged.
* Use of class III antiarrhythmics drugs (eg, dofetilide, ibutilide, amiodarone, bretylium, sotalol) within 30 days prior to TKR.

General

* Participation in any investigational drug study 30 days prior to enrollment is prohibited. Participation in a device trial prior to enrollment is acceptable.
* Any condition which could interfere with or for which the treatment of might interfere with the conduct of the study, or which would, in the opinion of the Investigator, unacceptably increase the risk of the subject's participation in the study. This would include, but is not limited to alcoholism, drug dependency or abuse, psychiatric disease, epilepsy or any unexplained blackouts.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2006-05; Primary Completion 2007-01 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 10 May 2006 and 12 February 2007, 215 patients were enrolled. After undergoing unilateral total knee replacement surgery, patients were randomized to 1 of 3 treatment groups (2:2:1 allocation). The study was open-label for randomization to enoxaparin versus betrixaban, but the 15 mg versus 40 mg dose of betrixaban was double-blind.
Pre-assignment Details: Patients scheduled to undergo elective primary unilateral total knee replacement (TKR) surgery were evaluated for eligibility 1 to 30 days before surgery (Screening). Consenting subjects who remained eligible for the study after TKR were randomized. 215 patients were randomized and all but 1 received at least 1 dose of study drug.
Period: Overall Study
Arm/Group | Betrixaban 15 mg | Betrixaban 40 mg | Enoxaparin
Started | 88 | 84 | 43
Completed | 84 | 77 | 42
Not Completed | 4 | 7 | 1
Not completed — Did not receive treatment | 1 | 0 | 0
Not completed — Adverse Event | 0 | 3 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 4 | 0
Not completed — Neurologist Wanted Pt to start Plavix | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized patients who took at least 1 dose of study medication after randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Betrixaban 15 mg | Betrixaban 40 mg | Enoxaparin | Total
Number analyzed (Participants) | 87 | 84 | 43 | 214
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (7.2) | 65.0 (7.9) | 61.9 (9.6) | 63.7 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 52 | 22 | 129
  Male | 32 | 32 | 21 | 85

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adjudicated Venous Thromboembolism (VTE)
Description: Incidence of adjudicated venous thromboembolism (VTE) through Day 10-14 following TKR where VTE is defined as DVT (proximal and/or distal) and/or PE. Patients were evaluated for VTE daily while hospitalized and were contacted every 2 to 4 days after discharge and before the day of the mandatory venogram to monitor for study endpoints
Time Frame: Through Day 10-14 following TKR surgery, at time of mandatory venogram
Population: All randomized patients who took at least 1 dose of study medication after randomization and for whom an evaluable venogram was available
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Betrixaban 15 mg | Betrixaban 40 mg | Enoxaparin
Number analyzed (Participants) | 70 | 65 | 40
Percentage of Participants | 20 [11.4 to 31.3] | 15.4 [7.6 to 26.5] | 10 [2.8 to 23.7]

2. Primary Outcome: Incidence of Adjudicated Overt Bleeding Events: Primary Safety Endpoint
Description: The incidence of adjudicated major and clinical relevant non-major bleeding. Major bleeding was defined as fatal, involving vital organs, requiring additional surgery or a new therapeutic procedure, or a bleeding index >=2. Bleeding Index was defined as the number of units of packed red blood cells or whole blood transfused plus the haemoglobin values before the bleeding episode minus the haemoglobin values after the bleed had stabilized (in g/dL)
Time Frame: Through follow-up at approximately 6 (±2) weeks after TKR surgery
Population: All randomized patients who took at least 1 dose of study medication after randomization.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Betrixaban 15 mg | Betrixaban 40 mg | Enoxaparin
Number analyzed (Participants) | 87 | 84 | 43
Percentage of Participants | 0 [0 to 4.2] | 2.4 [0.3 to 8.3] | 7.0 [1.5 to 19.1]

3. Secondary Outcome: Incidence of Adjudicated Pulmonary Embolism (PE) and All Deep Vein Thrombosis (DVT) (Proximal and Distal)
Description: Incidence of adjudicated pulmonary embolism (PE) and all deep vein thrombosis (DVT) (proximal and distal) through the time of venography on Day 10 to 14 and at follow-up at approximately 6 (±2) weeks after TKR surgery
Time Frame: At follow-up at approximately 6 (±2) weeks after TKR surgery
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Betrixaban 15 mg | Betrixaban 40 mg | Enoxaparin
Number analyzed (Participants) | 70 | 65 | 40
Percentage of Participants | 20 [11.4 to 31.3] | 15.4 [7.6 to 26.5] | 12.5 [4.2 to 26.8]

ADVERSE EVENTS:
Time Frame: Through follow-up at approximately 6 (±2) weeks after TKR surgery
Description: Serious adverse events by system organ class
Arm/Group | Betrixaban 15 mg | Betrixaban 40 mg | Enoxaparin
Serious Adverse Events (participants affected / at risk) | 3/87 | 6/84 | 1/43
Other Adverse Events (participants affected / at risk) | 83/87 | 80/84 | 29/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Betrixaban 15 mg (N=87) | Betrixaban 40 mg (N=84) | Enoxaparin (N=43)
Sepsis (Infections and infestations) | 1 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0
Acute renal failure (Renal and urinary disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Betrixaban 15 mg (N=87) | Betrixaban 40 mg (N=84) | Enoxaparin (N=43)
Procedural pain (Injury, poisoning and procedural complications) | 52 | 43 | 3
Nausea (Gastrointestinal disorders) | 32 | 38 | 7
Constipation (Gastrointestinal disorders) | 26 | 18 | 8
Body temperature (Investigations) | 16 | 16 | 8
Vomiting (Gastrointestinal disorders) | 12 | 13 | 1
Pyrexia (General disorders) | 6 | 13 | 3
OEDEMA PERIPHERAL (General disorders) | 5 | 11 | 4
HYPOKALAEMIA (Metabolism and nutrition disorders) | 9 | 10 | 1
ANAEMIA (Blood and lymphatic system disorders) | 8 | 9 | 1
HYPOTENSION (Vascular disorders) | 6 | 8 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 10 | 6 | 0
HAEMOGLOBIN DECREASED (Investigations) | 5 | 6 | 3
POSTOPERATIVE FEVER (Injury, poisoning and procedural complications) | 8 | 5 | 3
INSOMNIA (Psychiatric disorders) | 14 | 4 | 5
DYSPEPSIA (Gastrointestinal disorders) | 5 | 4 | 0
RESPIRATORY GAS EXCHANGE DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0
LOCAL SWELLING (General disorders) | 9 | 3 | 1
DIZZINESS (Nervous system disorders) | 5 | 3 | 2
BLOOD POTASSIUM DECREASED (Investigations) | 2 | 3 | 2
WOUND SECRETION (Injury, poisoning and procedural complications) | 2 | 3 | 2
RASH (Skin and subcutaneous tissue disorders) | 1 | 3 | 2
DIARRHOEA (Gastrointestinal disorders) | 1 | 3 | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1
SINUS TACHYCARDIA (Cardiac disorders) | 1 | 3 | 0
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 0 | 3 | 0
INCISION SITE ERYTHEMA (Injury, poisoning and procedural complications) | 0 | 3 | 0
RALES (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 1
PROCEDURAL NAUSEA (Injury, poisoning and procedural complications) | 6 | 1 | 1
HEADACHE (Nervous system disorders) | 3 | 1 | 2
BREATH SOUNDS ABNORMAL (Investigations) | 3 | 1 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 | 1 | 3
ANXIETY (Psychiatric disorders) | 2 | 1 | 2
OXYGEN SATURATION DECREASED (Investigations) | 4 | 0 | 0
BLISTER (Skin and subcutaneous tissue disorders) | 3 | 0 | 1
ERYTHEMA (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
PLATELET COUNT INCREASED (Investigations) | 0 | 0 | 3
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Due to multiple studies, centers and countries this will vary.